CLINICAL TRIAL: NCT03153995
Title: Alveolar Ridge Augmentation Following Self-Inflating Soft Tissue Expander: A Randomized Controlled Clinical and Histological Study
Brief Title: Alveolar Ridge Augmentation Following Self-Inflating Soft Tissue Expander
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Talaat Ali, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-REC per-16-3
Record Dates: First submitted 2017-05-04; First posted 2017-05-15 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Horizontal Ridge Deficiency
Keywords: expander

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sub-periosteal soft tissue expansion (Experimental): Eight patients will receive osmotic hydrogel expanders prior to bone augmentation procedures. All expanders will be placed in sub-periosteal positions using the tunnel technique.
  Interventions: Procedure: soft tissue expansion
- periosteal releasing incision (Active Comparator): periosteal releasing incision will be performed for Eight patients during ridge augmentation surgery .
  Interventions: Procedure: soft tissue expansion

INTERVENTIONS:
Procedure: soft tissue expansion — Three surgeries will be carried out for group I patients:
  * Soft tissue expansion (1st surgery); at baseline
  * Alveolar ridge augmentation (2nd surgery); after five weeks
  * Implant surgery (3rd surgery); after six months
  Other Names: osmed

SUMMARY:
The objective of this study will be to assess and compare between sub-periosteal self- inflating osmotic tissue expanders used as preparatory surgery before alveolar ridge augmentation and periosteal releasing incision using autogenous onlay block bone graft.

The assessment and comparison will be based on:

1. Change in edentulous alveolar ridge in bucco-lingual dimension after alveolar

   ridge augmentation.
2. Quantity of the soft tissue obtained after soft tissue expansion.

DETAILED DESCRIPTION:
* Sixteen patients will be selected from the outpatient clinic of the department of, Oral medicine Periodontology, and oral diagnosis, Faculty of Dentistry, Ain Shams University.
* Three surgeries will be carried out for group I patient; the first is placement of soft tissue expander, the second surgery is bone grafting and placement of collagen membrane for ridge augmentation while the third (re-entry surgery) is implant placement in a routine fashion.

two surgeries will be carried out for group II patient; the first is surgery is bone grafting for ridge augmentation while the second (re-entry surgery) is implant placement in a routine fashion.

-Measurements and evaluation of edentulous ridge will be done by CBCT

ELIGIBILITY:
Inclusion Criteria:

* All patients should have partially edentulous ridge (missing upper one or two neighboring anterior teeth or premolars) of the maxilla. The edentulous area should require horizontal bone augmentation procedures owing to lack of sufficient residual bone.
* All patients should not have any particular medical history (medically free) according to Burket health medical history questionnaire (Glick et al.2008).
* All patients should not have any known contraindication to oral surgery.

Exclusion Criteria:

* Smokers will be excluded from our study.
* Patients with poor oral hygiene or not willing to perform oral hygiene measures.
* Patients who showed residual infections in the edentulous area or apparent infection in a neighboring tooth.
* Patients with systemic diseases such as diabetes mellitus and hemorrhagic disorders, patients receiving intravenous bisphosphonate therapy or systemic corticosteroid treatment.
* Patients with occlusal discrepancies will be excluded.
* Vulnerable groups (as pregnant and lactating females, and decisionaly impaired individuals) will be excluded from the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in ridge dimensional alteration by CBCT | baseline, 6 months after surgery, 3 months after implant surgery
  The ridge width will be compared between the two treatment groups by CBCT

SECONDARY OUTCOMES:
Soft tissue volume gain | baseline, 4 weeks
  Soft tissue volume gain will be assessed by volumetric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Amr, lecturer, Study Director — Ainshams University; Nevine Kheir eldin, professor, Study Director — Ainshams University; Ehab Abd elhamid, professor, Study Director — Ainshams University
Locations (1):
- Faculty of dentistry Ain Shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No